CLINICAL TRIAL: NCT00383318
Title: Demographic, Metabolic, and Genomic Description of Neonates With Severe Hyperbilirubinemia
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Other Study IDs: PDX 06-001
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Hyperbilirubinemia; Jaundice
Keywords: Neonate; Hyperbilirubinemia; Jaundice; G6PD Deficiency; Gilbert's Syndrome
MeSH Terms: conditions — Hyperbilirubinemia; Jaundice; Glucosephosphate Dehydrogenase Deficiency; Gilbert Disease

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Gene mutation sample

SUMMARY:
The purpose of this study is to compare the demographic, metabolic, and genomic characteristics of patients who develop severe hyperbilirubinemia to patients who never developed a significant bilirubin level.

DETAILED DESCRIPTION:
The purpose of this study is to compare the demographic, metabolic, and genomic characteristics of patients who develop severe hyperbilirubinemia (serum bilirubin level in the "high risk zone of greater than the 95th percentile based on the Bhutani nomogram) to patients who never developed significant hyperbilirubinemia (bilirubin level in "low risk zone of less than the 40th percentile" on Bhutani nomogram and who did not require any treatment for hyperbilirubinemia). Our primary goal is to determine if common gene mutations occur at a greater frequency in patients with severe hyperbilirubinemia than in neonates without significant hyperbilirubinemia.

The gene mutations we will test for are:

* Glucose-6-phosphate Dehydrogenase Deficiency [G6PD] gene mutations
* African A- mutation (G202A;A376G)
* The common Mediterranean mutation (C563T)
* Two common Chinese mutations (G1376T and G1388A)
* UGT1A1 polymorphism. The UGT1A1 gene polymorphisms refer to those genetic defects found to be associated with Gilbert's Syndrome, including a promoter defect (T-3263G) that disrupts a transcription regulatory site, the TA repeats promoter polymorphism, and four mutations within the coding region (G211A, C686A, C1091T, and T1456G).
* Gene polymorphism for the organic anion transporting protein (OATP-2)

ELIGIBILITY:
Inclusion Criteria:

Case

* Documentation of informed consent.
* Gestational age greater than or equal to 37 weeks.
* Birth weight greater than or equal to 2000 grams.
* At least one serum bilirubin level that is greater than the 95th percentile ("high risk zone") based on the Bhutani nomogram(1), for the case population.
* Age at enrollment less than 7 days or less than or equal to 168 hours.
* No major anomalies (chromosomal abnormalities, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia, or other major gastrointestinal anomalies, major neurological injury or anomaly, and multiple congenital anomalies).
* Ability to follow subjects transferred to another facility for outcome data.

Control

* Documentation of informed consent.
* Gestational age greater than or equal to 37 weeks.
* Birth weight greater than or equal to 2000 grams.
* At least one estimate of serum bilirubin. Bilirubin level estimated to be less than the 40th percentile ("low risk zone") based on the Bhutani nomogram. While a serum bilirubin in the low risk zone is the preferred method for assessing the bilirubin level, many pediatricians use transcutaneous measure of bilirubin as a screening tool for identifying "low risk" patients. For this reason, we will allow controls to be identified using transcutaneous measurements and collect serum bilirubin levels only as clinically indicated.
* Age at enrollment less than 7 days or less than or equal to 168 hours.
* No major anomalies (chromosomal abnormalities, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia or other major gastrointestinal anomalies, major neurological injury or anomaly, and multiple congenital anomalies).
* Ability to follow subjects transferred to another facility for outcome data.

Exclusion Criteria:

Case and Control

* Gestational age less than 37 weeks.
* Birth weight less than 2000 grams.
* Older than 7 days of age or 168 hours.
* Any major congenital anomalies.

Max Age: 6 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reese H Clark, MD, Principal Investigator — Pediatrix; Zhili Lin, PhD, MD, Principal Investigator — Pediatrix Screening; Jon Watchko, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Greenville Medical Center, Greenville, South Carolina, United States

REFERENCES:
- [Background] Watchko JF. Vigintiphobia revisited. Pediatrics. 2005 Jun;115(6):1747-53. doi: 10.1542/peds.2004-1748. PMID 15930239
- [Background] Bhutani VK, Johnson LH, Jeffrey Maisels M, Newman TB, Phibbs C, Stark AR, Yeargin-Allsopp M. Kernicterus: epidemiological strategies for its prevention through systems-based approaches. J Perinatol. 2004 Oct;24(10):650-62. doi: 10.1038/sj.jp.7211152. PMID 15254556
- [Background] Johnson LH, Bhutani VK, Brown AK. System-based approach to management of neonatal jaundice and prevention of kernicterus. J Pediatr. 2002 Apr;140(4):396-403. doi: 10.1067/mpd.2002.123098. No abstract available. PMID 12006952
- [Background] Ip S, Chung M, Kulig J, O'Brien R, Sege R, Glicken S, Maisels MJ, Lau J; American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. An evidence-based review of important issues concerning neonatal hyperbilirubinemia. Pediatrics. 2004 Jul;114(1):e130-53. doi: 10.1542/peds.114.1.e130. PMID 15231986
- [Derived] Watchko JF, Lin Z, Clark RH, Kelleher AS, Walker MW, Spitzer AR; Pediatrix Hyperbilirubinemia Study Group. Complex multifactorial nature of significant hyperbilirubinemia in neonates. Pediatrics. 2009 Nov;124(5):e868-77. doi: 10.1542/peds.2009-0460. Epub 2009 Oct 26. PMID 19858149